CLINICAL TRIAL: NCT01528956
Title: Using New Approaches for Genomics Studies in Pediatric Adrenocortical Tumors: Whole Genome Sequencing; Deep Sequencing; miRNA; methDNA and SNP 6.0
Brief Title: Studying Genes in Samples From Younger Patients With Adrenocortical Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ARAR12B1; COG-ARAR12B1 (Other: Children's Oncology Group); CDR0000724572 (Other: Clinical trials.gov); ARAR12B1 (Other: Children's Oncology Group); NCI-2012-00244 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-05; First posted 2012-02-08 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Adrenocortical Carcinoma
Keywords: adrenocortical carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — DNA Methylation; Gene Expression Profiling; Base Sequence; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: nucleic acid sequencing
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of blood and tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies genes in samples from younger patients with adrenocortical tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To perform whole-genome sequencing, deep sequencing, micro RNA analysis, methylation status, copy number variation analysis, and single-nucleotide polymorphisms (SNPs) analysis in pediatric adrenocortical tumors and compare those results to those of the same patient's normal cells.

OUTLINE: Archived tumor and blood samples are analyzed for whole-genome sequencing, deep sequencing, micro RNA , methylation status, copy variation, and single-nucleotide polymorphisms. Results are then compared with patients' normal cells.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Banked tumor and blood samples obtained from patients enrolled on COG-ARAR0332 in North America and Brazil

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients enrolled on COG-ARAR0332
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification of genetic factors affecting adrenocortical tumors
Comprehensive catalog of altered genes in adrenocortical samples

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Zambetti, PhD, Principal Investigator — St. Jude Children's Research Hospital